CLINICAL TRIAL: NCT06772259
Title: Comparison of the Effect of Two Different Interventions on Pain and Fear in Peripheric Intravenous Catheterization in Children: a Randomized Controlled Study
Brief Title: Comparison of the Effect of Two Different Interventions
Acronym: PIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: Sakarya University Education and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Ramazan BOZKURT, RN, MSc, PhD Candidate, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-16214662-050.01.04-236416-36
Record Dates: First submitted 2024-12-24; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: To Compare the Effect of Two Different Nonpharmacological Methods on Pain and Fear During Peripheral Intravenous Catheterization
Keywords: pain; fear; children; distraction; palm stimulator; cartoon; peripheral intravenous; catheterization; cannulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Palm stimulator group (Experimental): The Palm Stimulator is grasped in the palm during painful interventions and provides stimulation. Blunt protrusions around the apparatus provide tactile stimulation in the palm. The blunt protrusions have been found to reduce the pain perceived during the intervention by closing the pain gate in the spinal cortex by creating stimuli according to the gate control pain theory without penetrating the skin. The researchers who developed the apparatus were contacted via e-mail and permission was obtained for using the palm stimulator.
  In the study, the child held the palm stimulator in the palm during the PIK procedure, and the researcher evaluated pain and fear. After the PIK procedure was completed, the child was asked to release the apparatus from the palm.
  Interventions: Device: Palm Stimulator
- Cartoon group (Experimental): Distraction by watching cartoons is a promising, cost-effective, and non-pharmacologic technique to reduce pain in children undergoing painful procedures. The cartoon was selected by expert researchers from the pediatric field in the research team following the age and consciousness level of the children. A projection device was placed in the intervention room for data collection. The cartoon was projected on a blank wall in the intervention room. The cartoon was played in preparation for the PIK procedure, and children were allowed to watch it until it was completed.
  Interventions: Other: Cartoon
- Control gruup (No Intervention): In the control group, the routine application phase was performed. Age-appropriate children were seated in the blood sampling chair, and those who could not sit were placed on a stretcher, and PIK was performed. The parent was also taken to the intervention room during the procedure.

INTERVENTIONS:
Device: Palm Stimulator — The apparatus is 1.6 cm in diameter and 4 cm long. It has a cylindrical, non-slippery and easy-to-grasp structure for maximum contact with the palm
  Arms: Palm stimulator group
Other: Cartoon — The cartoon was projected on a blank wall in the intervention room with a projection device. The cartoon was played in preparation for the PIK procedure and children were allowed to watch it until the procedure was completed.
  Arms: Cartoon group

SUMMARY:
The goal of this clinical trial is to compare the effect of two different non-pharmacologic interventions with the control group in reducing pain due to peripheral intravenous catheterization application in children aged 5-12 years.

Hypotheses:

H1: Pain level differs in the group that received PIK with Palm Stimulator compared to the control group.

H2: The level of fear in the group with PIK application with Palm Stimulator differs from the control group.

H3: Satisfaction level is different in the group with PIK application with Palm Stimulator compared to the control group.

H4: The pain level differs in the group that received PIK application by watching cartoons compared to the control group.

H5: The level of fear is different in the group that received PIK application by watching cartoons compared to the control group.

H6: Satisfaction level is different in the group that received PIK application by watching cartoons compared to the control group.

H7: Pain level is different in the Palm Stimulator PIK group compared to the cartoon group.

H8: The level of fear is different in the Palm Stimulator PIK group compared to the cartoon group.

H9: The satisfaction level in the group with PIK application with Palm Stimulator is different from the cartoon group.

H10: PIK application time is different in the palm stimulator group compared to the control group.

H11: PIK application time is different in the cartoon group compared to the co

DETAILED DESCRIPTION:
1. To measure the pain and fear levels of children by placing a palm stimulator on their palms during PIK application
2. Measuring pain and fear levels by watching cartoons to children during PIK application

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the study,
2. Pediatric patients for whom written and verbal consent has been obtained from the parent,
3. Pediatric patients for whom verbal consent was obtained,

(3) Not under the influence of sedative/anticonvulsant/analgesic drugs, (4) Pediatric patients aged 5-12 years, (5) Pediatric patients who can communicate, understand, and carry out commands and are not dependent on technological devices.

Exclusion Criteria:

1. Not volunteering to participate in the study,
2. More than one PIK attempt,
3. Children with a chronic, acute, or life-threatening illness.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Pain Measurement | 3 months
  Before, during, and after the PIK procedure in intervention and control groups. Wong-Baker FACES Pain Scale: The scale used to diagnose pain in children was developed by Donna Lee Wong and Connie Morain Baker. The Wong-Baker Scale has been reported to be safe to use in children aged 3-18 who can verbally describe the level of pain. The scale includes facial expressions and numbers. The scale has a total of six facial expressions, and pain is graded between 0-10 (Wong & Baker, 1988).
Fear | 3 months
  Fear assessment before, during, and after the PIK procedure in intervention and control groups.
  Child Fear Scale: The Turkish psychometric properties of the scale adapted to pediatric patients as "Children's Fear Scale" by McMurty et al. (2011) were evaluated by Özalp Gerçeker et al. The CSA is a scale consisting of five drawn facial expressions ranging from neutral expression (0=no anxiety) to frightened face (4=severe anxiety) and evaluated between 0 and 4 (Özalp Gerçeker et al., 2018). It can be used by families and researchers to assess pain and anxiety before and during the procedure and is intended for children aged 5-10 years. In the Turkish reliability and validity study, the content validity index of the scale was found to be 0.89 (Özalp Gerçeker et al., 2018).

SECONDARY OUTCOMES:
Saticfaction | 3 months
  Satisfaction assessment after the PIK procedure in intervention and control groups.
  Individuals were asked to give a score between 0-10 to determine their satisfaction. A score of "0" means "not at all satisfied", while a score of "10" means "very satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scupola A, Tiberti AC, Sasso P, Mastrocola A, Berarducci A, Bozzoni Pantaleoni F, Da Dalt S, Balestrazzi E. SD-OCT imaging of idiopathic macular holes with spontaneous closure. Ophthalmic Surg Lasers Imaging. 2012 Feb 23;43 Online:e14-7. doi: 10.3928/15428877-20120216-01. PMID 22356437
- [Background] Suman Kc S, Sharma P, Singh H, Bal C, Kumar R. Fibrous Dysplasia Mimicking Bone Metastasis on Both Bone Scintigraphy and (18)F-FDG PET-CT: Diagnostic Dilemma in a Patient with Breast Cancer. Nucl Med Mol Imaging. 2012 Dec;46(4):318-9. doi: 10.1007/s13139-012-0171-7. Epub 2012 Sep 15. No abstract available. PMID 24900084
- [Background] Shaik JA, Guram G. A Comparative Evaluation of Canine Retraction Using Ceramic Bracket and Ceramic Bracket with Metal Slot with Conventional Preadjusted Edgewise Appliance Bracket Systems: A Clinical Study. J Int Soc Prev Community Dent. 2018 Jul-Aug;8(4):296-303. doi: 10.4103/jispcd.JISPCD_301_17. Epub 2018 Jul 18. PMID 30123760
- [Background] Otulakowski G, Kavanagh BP. Hydrogen sulfide in lung injury: therapeutic hope from a toxic gas? Anesthesiology. 2010 Jul;113(1):4-6. doi: 10.1097/ALN.0b013e3181dec00e. No abstract available. PMID 20574223
- [Derived] Bozkurt R, Dogu O, Arsoy HEM, Ozdemir O. Comparing Nonpharmacological Interventions for Pain, Fear, and Satisfaction: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Oct 1:S1524-9042(25)00275-9. doi: 10.1016/j.pmn.2025.09.004. Online ahead of print. PMID 41038771